CLINICAL TRIAL: NCT06824974
Title: Feasibility Study of Time Restricted Eating and a Healthy Diet in Patients Receiving Liver-Directed Therapy for Hepatocellular Carcinoma
Brief Title: To Test Whether Time-restricted Eating Coupled With a Healthy Diet is Beneficial in Liver Cancer Patients
Acronym: TRE+HE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Nicholas Webster, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: #808859
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Liver Cancer, Adult; MASH - Metabolic Dysfunction-Associated Steatohepatitis; Obesity and Overweight
Keywords: Time-restricted eating; healthy diet
MeSH Terms: conditions — Carcinoma, Hepatocellular; Obesity; Overweight; Intermittent Fasting | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will follow time-restricted consumption of a healthy diet.
  Interventions: Behavioral: Time-restricted eating plus healthy diet
- Control (No Intervention): Control observational arm.

INTERVENTIONS:
Behavioral: Time-restricted eating plus healthy diet — Subjects will restrict calorie consumption to 8-10 hours during the day plus will follow a healthy plant-based diet.
  Arms: Intervention

SUMMARY:
This is a feasibility study that will collect data to assess the potential effect of a nutritional intervention designed to improve liver metabolism. This prospective single-site trial will enroll adult patients undergoing liver-directed therapies for hepatocellular carcinoma. Eligible individuals who are randomized to the intervention group will be enrolled in a six-month nutritional change program consisting of time-restricted eating in which calorie consumption is limited to 8-10 hours during the day, plus targeted healthy changes in what they eat. The intervention includes dietary counseling visits with a study registered dietitian and motivational phone calls with a study Certified Health and Wellness Coach to help subjects adhere to the intervention. Individuals in the control group will be enrolled in a six-month period of observation only. The main questions it aims to answer are:

Is a prolonged nightly fast coupled with a healthy diet safe and feasible for patients with liver cancer? Does the intervention improve liver metabolism?

ELIGIBILITY:
Inclusion Criteria:

1. Overweight or obese (BMI 27-45 kg/m2)
2. BCLC early to intermediate stage HCC
3. Referred for liver-directed therapy (PTA, TACE, TARE within 3 months)
4. English or Spanish speaking over the age of 18.
5. ECOG Performance Status ≤ 2.
6. Usual nightly fasting <12 hours
7. Willing to comply with all study procedures
8. Child-Pugh A liver function.

Exclusion Criteria:

1. Advanced HCC, progression, and/or associated comorbidities, metastatic disease, tumor in vein, or ascites
2. Advanced Cirrhosis (hypoalbuminemia/Child-Pugh B+C). Poorly controlled or refractory (grade 3-4) hepatic encephalopathy
3. Type 1 diabetes or self-reported hypoglycemia or hypoglycemic events by CGM
4. Participation in another conflicting study that requires modification of diet or food timing.
5. Uncontrollable eating pattern (e.g., wasting, Night Eating Syndrome, disordered eating habits, food insecurity)
6. Medications that markedly impact metabolic study biomarkers.
7. Other cancer in last 10 years (other than nonmelanoma skin cancer or carcinoma of the cervix in situ)
8. Serious medical conditions such as chronic kidney disease, congestive heart failure, or any condition that would interfere with participation in the trial.
9. Unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy
10. Active alcohol abuse or less than 6 months of sobriety
11. Participation in a trial of an investigational agent within the prior 30 days
12. Pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to protocol | 6 months
  Participant adherence to and comprehension of the protocol as an indicator of intervention delivery by staff. Adherence will be assessed by the number of participants who complete the study, the percentage of days with fasting >14 h, and the number of days that food was logged into the app.
Safety from adverse events | 6 months
  Safety assessed by adverse events and liver function tests. Reports on adverse events will include hypoglycemic epidoes, nausea, disrupted sleep, decreased quality of life or other patient reported events from surveys. Liver function tests (AST and ALT) as well ss platelet count and total protein are monitored under SOC. AST and ALT elevation will be considered mild if 2-5 times upper limit normal (ULN), moderate if 5-15 times ULN, and severe if >15 times ULN.
Ability to recruit | 6 months
  Ability to recruit our target population will be assessed by the number of eligible individuals in the patient population, and the number who enroll in the trial.
Satisfaction and self-motivation | 6 months
  We will determine the degree to which participants liked the intervention through satisfaction surveys at the end of the study and the number of participants who demonstrate self-motivation to continue the intervention protocol during 6-month follow-up.

SECONDARY OUTCOMES:
Effect of intervention on Quality of Life | 6 months
  Quality of Life will be assessed using the EORTC QLQ C-30 questionnaire for Cancer patients
Effect of interventions on fasting glucose | 6-months
  Fasting glucose will be measured at baseline and 6 months
Sleep disturbance | 6 months
  Sleep disturbance as reported by the PROMIS-8b survey
Effect of intervention on body weight | 6 months
  Body weight will be measured prior to and during intervention
Effect of intervention on food frequency | 6 months
  Participants will complete a Food frequency questionnaire at Baseline, 3 months and 6 months
Effect of intervention on Adiposity | 6 months
  Adiposity will be measured by Dual-energy X-ray Absorptiometry (DXA) at baseline and at 6 months
Effect of interventions on Physical activity | 6 months
  Physical activity will be measured by Accelerometer mounted at the waist at baseline and at 6 months
Effect of intervention on Glucose levels | 6 months
  Glucose levels will be monitored by Continuous Glucose Monitoring at baseline and at 6 months
Effect of intervention on fasting insulin | 6 months
  Fasting insulin levels will be measured at baseline and at 6 months
Effect of intervention on ketone production | 6 months
  Fasting beta-hydroxybutyrate levels will be measured at baseline and 6 months
Effect of interventions on hemoglobin A1c | 6 months
  Hemoglobin A1c will be measured at baseline and 6 months
Effect of intervention on plasma leptin | 6 months
  Leptin levels will be measured at baseline and 6 months
Effect of intervention on inflammatory cytokines | 6 months
  Inflammatory cytokines will be measured at baseline and 6 months
Effect of intervention on fecal microbiome | 6 months
  7S sequencing will be performed on fecal samples at baseline and 6 months

OTHER OUTCOMES:
Disease progression as a Tertiary/Exploratory outcome | 12-months
  Tumor regression or recurrence will be assessed using LI-RADS-TR.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Webster, PhD, Principal Investigator — Universoty of California San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das M, Kumar D, Sauceda C, Oberg A, Ellies LG, Zeng L, Jih LJ, Newton IG, Webster NJG. Time-Restricted Feeding Attenuates Metabolic Dysfunction-Associated Steatohepatitis and Hepatocellular Carcinoma in Obese Male Mice. Cancers (Basel). 2024 Apr 16;16(8):1513. doi: 10.3390/cancers16081513. PMID 38672595
- [Background] Das M, Webster NJG. Obesity, cancer risk, and time-restricted eating. Cancer Metastasis Rev. 2022 Sep;41(3):697-717. doi: 10.1007/s10555-022-10061-3. Epub 2022 Aug 19. PMID 35984550